CLINICAL TRIAL: NCT04017364
Title: Treatment of Coronary De-novo Stenosis by a Sirolimus Coated Balloon or a Paclitaxel Coated Balloon Catheter
Brief Title: Treatment of Coronary De-novo Stenosis by a Sirolimus Coated Balloon or a Paclitaxel Coated Balloon Catheter Malaysia
Acronym: SCBDNMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoRa GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI-DN-MALAYSIA
Record Dates: First submitted 2019-07-03; First posted 2019-07-12 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: drug coated balloon; Paclitaxel; sirolimus
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTCA of coronary de novo lesion PCB (Active Comparator): Predilatation of coronary de-novo stenosis followed by a SeQuent®Please or SeQuent®Please Neo balloon (paclitaxel 3.0 μg/mm²)
  Interventions: Device: PCB PTCA
- PTCA of coronary de novo lesion SCB (Experimental): Predilatation of coronary de-novo stenosis followed by a sirolimus coated SeQuent®SCB balloon (sirolimus 4.0 μg/mm²)
  Interventions: Device: SCB PTCA

INTERVENTIONS:
Device: PCB PTCA — Predilatation of coronary de-novo stenosis followed by a PCB
  Arms: PTCA of coronary de novo lesion PCB
Device: SCB PTCA — Predilatation of coronary de-novo stenosis followed by a SCB
  Arms: PTCA of coronary de novo lesion SCB

SUMMARY:
To examine the treatment of coronary de-novo stenosis with a sirolimus coated balloon versus a paclitaxel coated balloon

DETAILED DESCRIPTION:
To examine the treatment of coronary de-novo stenosis with a sirolimus coated balloon versus a paclitaxel coated balloon. Prospective, multicenter, randomized, single-blind, 70 patients. Experimental intervention: Predilatation of coronary de-novo stenosis followed by a sirolimus coated SeQuent®SCB balloon (sirolimus 4.0 μg/mm²). Control intervention: Predilatation of coronary de-novo stenosis followed by a SeQuent®Please or SeQuent®Please Neo balloon (paclitaxel 3.0 μg/mm²). Follow-up per patient: 30 days telephone call; 6 months angiographic + 12 months. clinical follow up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of stable or unstable angina or a positive functional study
* Patients with significant coronary de-novo stenosis (≥ 70% diameter stenosis or intermediate ≥ 50% to <70% diameter stenosis with positive functional test or symptom of ischemia)
* Successful lesion preparation (no flow-limiting dissection or a residual stenosis > 30%)

Exclusion Criteria:

* Acute myocardial infarction within the past 72 hours (STEMI or NSTEMI)
* Intolerance and / or allergy to Sirolimus
* Intolerance or allergy to Paclitaxel and/or the delivery matrix (main ingredient:

iopromide)

* Patients with an ejection fraction of < 30 %
* Reference vessel diameter (RVD) < 2.5 mm
* Contraindication for whichever necessary accompanying medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
late lumen loss in-segment | 6 months
  angiographic minimal lumen diameter in-segment at 6 months minus minimal lumen diameter at baseline

SECONDARY OUTCOMES:
Procedural success | 5 days
  combined endpoint of: < 30% final diameter stenosis, no flow-limiting dissection (type C or higher), TIMI III flow, and the absence of in-hospital MACE
MACE | at 6 and at 12 months
  combined endpoint of: cardiac death, target vessel myocardial infarction, and TLR target lesion revascularization in-hospital at 6 and at 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- Malaysia (6):
  - Sabah Heart Centre, Queen Elizabeth Hospital II, Kota Kinabalu
  - National Heart Institute, Kuala Lumpur
  - Cardio Vascular Sentral, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak Heart Centre, Kuching
  - Hospital Pulau Pinang, Pulau Pinang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ali RM, Abdul Kader MASK, Wan Ahmad WA, Ong TK, Liew HB, Omar AF, Mahmood Zuhdi AS, Nuruddin AA, Schnorr B, Scheller B. Treatment of Coronary Drug-Eluting Stent Restenosis by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2019 Mar 25;12(6):558-566. doi: 10.1016/j.jcin.2018.11.040. PMID 30898253
- [Derived] Ahmad WAW, Nuruddin AA, Abdul Kader MASK, Ong TK, Liew HB, Ali RM, Mahmood Zuhdi AS, Ismail MD, Yusof AKM, Schwenke C, Kutschera M, Scheller B. Treatment of Coronary De Novo Lesions by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2022 Apr 11;15(7):770-779. doi: 10.1016/j.jcin.2022.01.012. Epub 2022 Mar 16. PMID 35305906